CLINICAL TRIAL: NCT06484725
Title: Oncotype DX in BRCA-mutated Breast Cancer Patients: Our Experience. A Retrospective Observational Monocentric Study
Acronym: OnBRA
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rosa Di Micco, MD, MD, PhD, IRCCS San Raffaele
Other Study IDs: CET 175-2024
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Genetic Predisposition
Keywords: BRCA1; BRCA2; Genomic test
MeSH Terms: conditions — Breast Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Wild type patients: Patients with no mutations or VUS in Breast Cancer-related genes candidated to surgery as primary treatment and eligible for Oncotype DX assay.
  Interventions: Genetic: Oncotype DX assay
- VUS patients: Patients with VUS in Breast Cancer-related genes candidated to surgery as primary treatment and eligible for Oncotype DX assay.
  Interventions: Genetic: Oncotype DX assay
- Mutated patients: Patients with mutation in Breast Cancer-related genes candidated to surgery as primary treatment and eligible for Oncotype DX assay.
  Interventions: Genetic: Oncotype DX assay

INTERVENTIONS:
Genetic: Oncotype DX assay — Oncotype DX assay (Genomic Health, Inc, Redwood City, Calif) is a 21 gene panel developed to predict the risk of tumor recurrence in patients with ER-positive and human epidermal growth factor 2 (HER2)- negative breast cancer (BC); nowadays, this test represents a standard of care to guide adjuvant chemotherapy decision recommended in several guidelines. According to Oncotype DX Recurrent Score (RS)® a high RS shows a worse prognosis and predicts chemotherapy benefit in patients with ER-positive HER2-negative BC.

SUMMARY:
The study aims to evaluate the distribution of the Oncotype DX RS® genomic test in patients with ER-positive and HER2-negative breast cancer treated from January 2012 to December 2021, focusing on patients presenting germline mutations.

DETAILED DESCRIPTION:
In the past decades, genetic testing for cancer susceptibility has become essential in breast cancer (BC) management. Up to 10% of BC cases are associated with an inherited mutation in various genes, especially BRCA 1 and BRCA 2. Estrogen receptor (ER) positivity is observed in 22% on BRCA 1 and 77% of BRCA 2 mutation carrier; moreover, other genes are strongly related to ER-positive cancer.

Oncotype DX assay (Genomic Health, Inc, Redwood City, Calif) is a 21 gene panel developed to predict the risk of tumor recurrence in patients with ER-positive and human epidermal growth factor 2 (HER2)- negative BC; nowadays, this test represents a standard of care to guide adjuvant chemotherapy decision recommended in several guidelines. According to Oncotype DX Recurrent Score (RS)® a high RS shows a worse prognosis and predicts chemotherapy benefit in patients with ER-positive HER2-negative BC.

Combining Oncotype DX RS® with other risk factor elements, in particular germline mutations, could help to select patients who would benefit from an appropriate adjuvant therapy.

This retrospective observational study aims to evaluate Oncotype DX RS® distribution in ER-positive HER2-negative BC patients treated from January 2012 to December 2021, focusing on patients harboring mutation in BC-associated genes compared to the general population.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis at least 18 years
* Women who underwent breast surgery in OSR
* Patients with ER-positive, HER2-unamplified early-stage BC who underwent the Oncotype DX assay, according to the standard of care.

Exclusion Criteria:

* Male
* ER negative or HER2 amplified disease
* Patient s who did not undergo breast surgery in OSR
* Patient s who did not undergo the Oncotype Dx assay

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who underwent surgery as primary treatment and eligible for Oncotype DX assay.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Oncotype DX assay and RS® in participants. | 30 days after surgery.
  To evaluate the Oncotype DX RS® distribution in ER-positive early BC patients comparing patients with a deleterious germline mutation, patients with a VUS in BC-related genes and patients with no mutation.

SECONDARY OUTCOMES:
Oncotype DX assay and RS® in participants by menopausal or nodal status. | 30 days after surgery
  To evaluate Oncotype DX RS® distribution stratifying patients by menopausal or nodal status.
Distant or local recurrence. | Up to 10 years after surgery
  Evaluation of distant or local recurrence from follow-up data

CONTACTS AND LOCATIONS:
Overall Officials: Oreste Davide Gentilini, Study Director — Vita-Salute San Raffaele University
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No